CLINICAL TRIAL: NCT03792789
Title: Evaluation of Repetitive Transcranial Magnetic Stimulation as an Adjunct to Modified Constraint Induced Movement Therapy in Improving Upper Limb Function in Children With Hemiparetic Cerebral Palsy Aged 5 - 18 Years - A Randomized Controlled Trial
Brief Title: Evaluation of Repetitive Transcranial Magnetic Stimulation as an Adjunct to Modified Constraint Induced Movement Therapy in Improving Upper Limb Function in Children With Hemiparetic Cerebral Palsy Aged 5 - 18 Years
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Sheffali Gulati, Professor, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IECPG/574/11/2018
Record Dates: First submitted 2018-12-19; First posted 2019-01-03 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2019-01

CONDITIONS: Hemiparetic Cerebral Palsy
Keywords: Transcranial Magnetic Stimulation (TMS); modified Constraint Induced Movement Therapy (mCIMT)

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mCIMT with real rTMS (Experimental): Modified Constraint Induced Movement Therapy (mCIMT) with real Repetitive Transcranial Magnetic Stimulation (rTMS). 10 sessions of mCIMT will be administered using physical rehabilitation protocol along with real rTMS over contralateral primary motor cortex.
  Interventions: Device: mCIMT with real rTMS
- mCIMT with sham rTMS (Sham Comparator): Modified Constraint Induced Movement Therapy with sham Repetitive Transcranial Magnetic Stimulation (using sham coil). 10 sessions of mCIMT will be administered using physical rehabilitation protocol along with sham rTMS over contralateral primary motor cortex using sham coil which simulated sound and touch of real coil but has no electro-magnetic waves.
  Interventions: Device: mCIMT with sham rTMS

INTERVENTIONS:
Device: mCIMT with real rTMS — Modified constraint induced movement therapy will be provided to all children according to predefined protocol.
  rTMS will be provided using figure of eight shaped coil and TMS stimulator ((Magventure Denmark, X100 with mapoption) over contra-lesional primary motor cortex over 10 sessions of 20 minutes each spread over 4 weeks. Each session will comprise priming ( 10 minutes of 6Hz rTMS at 90% of resting motor threshold, delivered in two trains per minute with 5 seconds per train and 25-seconds intervals between trains (a total of 600 priming pulses)). Priming will be followed immediately by additional 10 minutes of 1Hz rTMS at 90% of resting motor threshold without interruption (a total of 600 low-frequency pulses).
  Arms: mCIMT with real rTMS
Device: mCIMT with sham rTMS — Modified constraint induced movement therapy will be provided to all children according to predefined protocol.
  Sham rTMS will be given using a sham coil.
  Arms: mCIMT with sham rTMS

SUMMARY:
The investigators aim to evaluate efficacy of TMS as an adjunct to CIMT, assess its safety and tolerability and study cortical excitability with help of TMS which are both rehabilitative therapies for hemiplegic cerebral palsy.

DETAILED DESCRIPTION:
Cerebral palsy is the most common motor disability of childhood and Hemiparetic cerebral palsy accounts for about one third of cases. Improving spasticity and upper limb function in these children can lead to better functional outcome and quality of life. TMS is an upcoming rehabilitative modality which has shown promising results in western studies. It has benefits of being non-invasive and has shown to have additive effect when used with CIMT which is standard of care in hemiparetic CP. However, randomized controlled clinical trials comparing it with CIMT alone in hemiparetic CP are very few, none from India so far. The dose, type and duration of TMS and its feasibility in resource limited set up needs to be investigated in children .Therefore, the investigators aim to evaluate efficacy of TMS as an adjunct to CIMT, assess its safety and tolerability and study cortical excitability with help of TMS.

ELIGIBILITY:
Inclusion Criteria:

* • Age 5 - 18 years

  * Hemiparetic Cerebral Palsy (perinatal brain injury)
  * Intelligence Quotient >70 (Binet Kamat Test/Malin's Intelligence Scale for Children)
  * Modified Ashworth scoring 1-3 for affected limb
  * Can sit independently or with support (GMFCS stage : 1-4 and Manual Ability Classification System stage: 1-3)
  * Preserved vision and hearing (with or without correction)

Exclusion Criteria:

* • Uncontrolled epilepsy as defined by seizure frequency >1/month for preceding 3 months

  * Severe concurrent illness or disease not associated with CP or unstable medical conditions like pneumonia
  * Genetic or syndromic associations
  * Children diagnosed with Autistic Spectrum Disorders
  * Modified Ashworth Scale Score more than 3 at shoulder/elbow/wrist
  * Contractures of affected limb
  * Severe movement disorder like dystonia, choreo-athetosis or ballismus interfering with purposeful limb movement
  * Any congenital brain malformation detected on conventional MRI brain
  * Recent surgery/cast/splint in affected limb
  * Botulinum toxin/phenol block in affected limb in past 6 months or planned to receive in study period
  * Those receiving tone modifying agents within two weeks before enrolment (Tizanidine, baclofen, benzodiazepines, dantrolene)
  * mCIMT received in last 6 months
  * Any contraindications for TMS - implanted electronic device and non-removable metallic objects near coil e.g. Pacemaker, cochlear implant

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-01-15 (Estimated); Primary Completion 2020-08-01 (Estimated); Study Completion 2020-08-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy of 4 weeks of mCIMT with sham/real rTMS | Within 1 week of end of 4 weeks of mCIMT with sham/real rTMS
  ◦ To evaluate the efficacy of repetitive Transcranial Magnetic Stimulation (rTMS) as an adjunct to modified Constraint Induced Movement Therapy (mCIMT) for 4 weeks in improving the Upper Limb Function as per increase in total QUEST score by 5 in 5-18 years old children with Hemiparetic Cerebral Palsy

SECONDARY OUTCOMES:
To evaluate improvement in dissociated movements, grasp, weight bearing and protective extension in each group at the end of 4 weeks | within 1 week of end of 4 weeks of mCIMT with sham/real rTMS
  To evaluate improvement in dissociated movements, grasp, weight bearing and protective extension in each group at the end of 4 weeks
To evaluate improvement in speed of upper limb movements in each group at the end of 4 weeks | within 1 week of end of 4 weeks of mCIMT with sham/real rTMS
  To evaluate improvement in speed of upper limb movements in each group at the end of 4 weeks
To evaluate improvement in muscle strength in each group at the end of 4 weeks | within 1 week of end of 4 weeks of mCIMT with sham/real rTMS
  To evaluate improvement in muscle strength in each group at the end of 4 weeks
To assess improvement in quality of life after the intervention in each group | within 1 week of end of 4 weeks of mCIMT with sham/real rTMS
  To assess improvement in quality of life after the intervention in each group
To assess compliance to therapy in each group by Daily Compliance Log | within 1 week of end of 4 weeks of mCIMT with sham/real rTMS
  To assess compliance to therapy in each group by Daily Compliance Log
To study for adverse events of TMS | within 1 week of end of 4 weeks of mCIMT with sham/real rTMS
  To study for adverse events of TMS
To evaluate cortical excitability with TMS at baseline and the end of 4 weeks | within 1 week of end of 4 weeks of mCIMT with sham/real rTMS
  To evaluate cortical excitability with TMS at baseline and the end of 4 weeks
• To evaluate sustenance of improvement by change in QUEST score at the end of 12 weeks, 8 weeks after stopping supervised treatment in both the groups | within 1 week of end of 4 weeks of mCIMT with sham/real rTMS
  • To evaluate sustenance of improvement by change in QUEST score at the end of 12 weeks, 8 weeks after stopping supervised treatment in both the groups

CONTACTS AND LOCATIONS:
Overall Officials: Sheffali Gulati, MD, Principal Investigator — All India Institute of Medical Sciences
Locations (1):
- India, New Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gupta J, Gulati S, Singh UP, Kumar A, Jauhari P, Chakrabarty B, Pandey RM, Bhatia R, Jain S, Srivastava A. Brain Stimulation and Constraint Induced Movement Therapy in Children With Unilateral Cerebral Palsy: A Randomized Controlled Trial. Neurorehabil Neural Repair. 2023 May;37(5):266-276. doi: 10.1177/15459683231174222. Epub 2023 May 11. PMID 37170480